CLINICAL TRIAL: NCT02064140
Title: Reducing High Respiratory Drive to Facilitate Supported Ventilation in ARDS Patients: a Pilot Study
Brief Title: Supported Ventilation in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Leo Heunks, L. Heunks, MD PhD, University Medical Center Nijmegen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MV NMBA JNLH13
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation; Tidal Volume
Keywords: ARDS; Mechanical Ventilation; Tidal volume; NMBA
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neuromuscular blocking agent (Experimental)
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium

SUMMARY:
Acute respiratory distress syndrome (ARDS) is characterized by acute bilateral pulmonary infiltrates and impairment of oxygen uptake. For example, pneumonia can cause the development of ARDS. Despite modern intensive care treatment, mortality in ARDS patients remains high (40%). Invasive mechanical ventilation (MV) is the mainstay of ARDS treatment. Controlled MV is the conventional ventilation strategy to ensure lung protective ventilation (low tidal volumes) and recovery of the lungs. However, among disadvantages of controlled MV are the development of respiratory muscle atrophy (due to disuse) and the need for high dose sedatives to prevent patient-ventilator asynchrony. The use of high doses of sedatives and respiratory muscle weakness are associated with increased morbidity, worse clinical outcomes and prolonged MV.

Besides controlled MV, a patient can be ventilated with supported ventilation. Supported MV decreases the likelihood to develop muscle atrophy, improves oxygenation and hemodynamics, and lowers consumption of sedatives. However potential disadvantages of supported ventilation include generation of too high tidal volumes, especially in patients with high respiratory drive. A previous study in healthy subjects has shown that titration of neuromuscular blocking agent (NMBA) can decrease activity of inspiratory muscles, while maintaining adequate ventilation. It is hypothesized that low dose NMBA may enable supported MV with adequate tidal volumes, in patients with high respiratory drive.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year
* informed consent
* ARDS according to the Berlin definition
* RASS -4/-5
* tidal volume > 8 ml/kg during supported ventilation
* double balloon esophageal EMG NAVA catheter

Exclusion Criteria:

* recent use of muscle relaxants / NMBAs (< 3 hours)
* pre-existent neuromuscular disease (congenital or acquired) or diseases / disorders know to be associated with myopathy including auto-immune diseases
* phrenic nerve lesions
* elevated intracranial pressure or clinical suspicion of elevated intracranial pressure (i.e. neurotrauma)
* open chest or abdomen
* pregnancy
* systolic blood pressure < 90 mm Hg / MAP < 65 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of titrating tidal volume < 6 ml/kg | Within 5 minutes after titration of NMBA
  The feasibility of titrating tidal volume in ARDS patients below 6 ml/kg using NMBA is evaluated in every patient. The outcome measure is dichotomic (yes/no).

SECONDARY OUTCOMES:
Respiratory rate | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA
  A secondary outcome measure is the respiratory rate after titration NMBA during different ventilatory modes.
Diaphragm electrical activity | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA.
  A secondary outcome measure is the root-mean-square of the diaphragm electrical activity after titration NMBA during different ventilatory modes.
Transpulmonary pressure | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA.
  Transpulmonary pressure is determined as the difference between mouth pressure and esophageal pressure during inspiration. Breath-by-breath data are ensemble-averaged over the first 2 minutes after titration NMBA during different ventilatory modes.
Transdiaphragmatic pressure | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA.
  Transdiaphragmatic pressure is determined as the difference between gastric pressure and esophageal pressure during inspiration. Breath-by-breath data are ensemble-averaged over the first two minutes after titration NMBA during different ventilatory modes.
Neuroventilatory efficiency | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA.
  A secondary outcome measure is the neuroventilatory efficiency (i.e. the ratio of diaphragm electrical activity and tidal volume) after titration NMBA during different ventilatory modes.
Neuromechanical efficiency | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA.
  A secondary outcome measure is the neuromechanical efficiency (i.e. the ratio of diaphragm electrical activity and transdiaphragmatic pressure) of the diaphragm after titration NMBA during different ventilatory modes.
Patient-ventilator contribution to breathing | During titration of NMBA (each three minutes) and during PS and NAVA after titration NMBA
  A secondary outcome measure is the patient-ventilator contribution to breathing (i.e. ratio of: the ratio of tidal volume and diaphragm electrical activity without assist, and the ratio of tidal volume and diaphragm electrical acticity with assist) during and after titration of NMBA.
Oxygenation index | Before start of the study; before titration of NMBA during different ventilatory modes; after titration of NMBA; after an hour for each ventilatory mode.
  A secondary parameter is the oxygenation index which is determined as the ratio between arterial oxygen tension and fraction of inspired oxygen.
Carbon dioxide tension in arterial blood (PaCO2) | Before start of the study; before titration of NMBA during different ventilatory modes; after titration of NMBA; after an hour for each ventilatory mode.
  A secondary parameter is the carbon dioxide tension in arterial blood.
pH of arterial blood | Before start of the study; before titration of NMBA during different ventilatory modes; after titration of NMBA; after an hour for each ventilatory mode.
  A secondary parameter is the pH of arterial blood.
Patient-ventilator interaction | Artefact-free period in the first 15 minutes during different ventilatory modes after titration of NMBA.
  Patient-ventilator interaction is evaluated using the NeuroSync index during different ventilatory modes.

CONTACTS AND LOCATIONS:
Overall Officials: L MA Heunks, MD, PhD, Principal Investigator — University Medical Center Nijmegen
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands